CLINICAL TRIAL: NCT05336435
Title: A Randomized Clinical Trial (RCT) of Population and Sex-specific Troponin Cutoffs for Ruling Out Acute Myocardial Infarction - The Danish Study of Population and Sex-Specific Cutoffs of Troponin
Brief Title: A Study of Population and Sex-specific Troponin Cutoffs for Ruling Out Acute Myocardial Infarction
Acronym: DANSPOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Nordsjaellands Hospital (Other); Amager Hospital (Other); Bispebjerg Hospital (Other); Zealand University Hospital (Other); Slagelse Sygehus (Other); Nykøbing Falster County Hospital (Other); Holbaek Sygehus (Other); Odense University Hospital (Other); Svendborg Hospital (Other); Kolding Sygehus (Other); Aarhus University Hospital (Other); Gødstrup Hospital (Other); Central Jutland Regional Hospital (Other); Randers Regional Hospital (Other); Glostrup University Hospital, Copenhagen (Other); Hvidovre University Hospital (Other); Vejle Hospital (Other); Hospital of Southern Jutland (Other); Horsens Hospital (Other); Aalborg University Hospital (Other); Regionshospital Nordjylland (Other Government); Sydvestjysk Sygehus (Unknown); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Professor, Consultant, DMSc, Herlev Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: FSP 20067240
Record Dates: First submitted 2022-03-29; First posted 2022-04-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Coronary Syndrome, Acute; Coronary Artery Disease; Myocardial Infarction
Keywords: coronary syndrome; myocardial infarction; clinical assessment; biomarker; troponin
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Intervention Model Description: A nationwide cluster-randomized trial with "stepped-wedge" design
Who Masked: Outcomes Assessor
Masking Description: A diagnosis of acute MI will be adjudicated for all individuals in the primary cohort by an endpoint committee consisting of three cardiologists from another region in Denmark.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm - Current sex-uniform manufacturer provided 99th percentile URL of troponin (No Intervention): Standard use of the current sex-uniform manufacturer provided 99th percentile URL of troponin is utilized at Danish hospitals as a diagnostic cutoff for acute MI for both men and women
- Intervention Arm - New population and sex-specific 99th percentile URLs of troponin (Active Comparator): Implementation of the new population and sex-specific 99th percentile URLs of troponin for the specific assay utilized at the enrolled centers.
  Interventions: Diagnostic Test: Implementation of the new population and sex-specific 99th percentile URL for cardiac troponin

INTERVENTIONS:
Diagnostic Test: Implementation of the new population and sex-specific 99th percentile URL for cardiac troponin — The new population and sex-specific 99th percentiles URLs will be implemented at all Danish hospitals receiving patients with chest pain for initial diagnostics for possible acute MI. This will take place as a randomized step-by-step introduction of population and sex-specific 99th percentile URLs for troponin in all hospital centers with a monthly start time interval. Each center is randomized to shifting from the sex-uniform manufacturer provided 99th percentile URL of cardiac troponin currently used nationwide to the new population and sex-specific 99th percentiles URLs provided by the DANSPOT study's first phase.
  Arms: Intervention Arm - New population and sex-specific 99th percentile URLs of troponin

SUMMARY:
Acute myocardial infarction (MI) is defined as a rise and/or fall in cardiac troponins (cTn) with at least one value above the 99th percentile upper reference limit (URL) in the context of symptoms or clinical evidence of myocardial ischemia. The URL is based on measurements in a healthy reference population. Currently, a sex-uniform manufacturer provided 99th percentile URL of troponin is utilized at Danish hospitals as a diagnostic cutoff for acute MI for both men and women. Reportedly, healthy men have twofold the troponin level compared to healthy women, suggesting that the use of a uniform URL for troponins may lead to the under-diagnostication of acute MI in women and potentially over-diagnostication in men.

The purpose of the DANSPOT study is to evaluate the clinical effect on diagnosis, treatment and outcomes in men and women presenting with acute MI of implementing international guidelines recommendations of sex-specific 99th percentile URLs for troponin into clinical practice.

First, to determine the sex-specific 99th percentile URLs of troponins based on a healthy Danish reference population, blood samples from Danish blood donors, were analyzed using one troponin T assay and four troponin I assays. Second, the DANSPOT study is a nationwide cluster-randomized trial with "stepped-wedge" design with participation of all 22 Danish hospital laboratories and associated departments of cardiology. With one-month intervals, each of 22 centers are randomized to shift from the presently applied uniform 99th percentile URL of troponin to our newly determined population and sex-specific 99th percentiles URLs. Each patient is followed in Danish registries for 12 months after first admission.

The hypothesis of the DANSPOT study is that implementation of population and sex-specific 99th URLs for troponin, will ensure that the right patients receive the right treatment. The investigators expect to detect significantly more women with acute MI, theoretically resulting in a more accurate diagnosis and treatment of women and men with acute MI.

DETAILED DESCRIPTION:
The present use of non-sex specific diagnostic cut-off levels of troponins in the diagnosis of acute myocardial infarction (MI) leads to under-diagnostication of acute MI in women and over-diagnostication in men. The purpose of this study is to document this through a randomized nationwide clinical implementation of population and sex-specific cut-off levels.

Coronary artery disease (CAD) is globally the leading cause of mortality for men and women. The latest consensus statement defines myocardial infarction as 1) a rise and/or fall in cardiac troponins with 2) at least one value above the 99th percentile upper reference limit (URL) in the context of 3) symptoms or clinical evidence of myocardial ischemia. Thus, levels of cardiac troponins play a key role in the diagnostic work-up in general. Currently, uniform manufacturer-provided URLs, defined by the 99th percentile of cardiac troponins in a healthy reference population, is applied in Danish hospitals as a diagnostic cut-off for acute MI for both men and women.

Lower levels of cardiac troponins are seen in healthy women as compared to healthy men, i.e. twice as high levels are seen in men. On this basis the clinical use of one uniform 99th percentile URL for cardiac troponins - i.e. applying the same diagnostic levels for men and women - may lead to a systematic under-diagnostication of acute MI in women and potentially an over-diagnostication of acute MI in men. Accordingly, the use of sex-specific 99th percentile URL of cardiac troponins are now recommended in recent guidelines by international cardiological societies, but this remains to be introduced in clinical practice.

The 99th percentile URLs for cardiac troponins currently used in Danish Hospitals are provided by the manufacturer of each specific assay based on blood samples from a healthy reference population collected by the manufacturer. Studies have shown that the 99th percentile value is dependent on patient sex as well as on the reference population selected and the definition for "healthy" used in these studies. It is well known that the 99th percentile URL should stem from a local reference population. This recommendation has never been implemented in Denmark.

The overall purpose of the study is to evaluate the clinical effect of implementing population and sex-specific 99th percentile URL for cardiac troponins in Denmark.

To determine the sex-specific 99th percentile URLs of troponins based on a healthy Danish reference population, blood samples from healthy Danish blood donors, were analyzed using one troponin T assay and four troponin I assays. Second, the DANSPOT study is a nationwide cluster-randomized trial with "stepped-wedge" design with participation of all 22 Danish hospital laboratories and associated departments of cardiology. With one-month intervals, each of 22 centers are randomized to shift from the presently applied uniform 99th percentile URL of troponin to our newly determined population and sex-specific 99th percentiles URLs. Each patient is followed in Danish registries for 12 months after first admission.

The clinical significance of sex-specific 99th percentile URLs of troponin is poorly investigated and for the same reason not yet implemented in Denmark or many other countries. The basic hypothesis of the DANSPOT study is that the implementation of population and sex-specific 99th URLs for troponin, will ensure that the right patients receive the right treatment. The investigators expect to detect significantly more women with acute MI, theoretically resulting in a more accurate diagnosis and treatment of women and men with acute MI. This would be guideline-defining for implementing sex-specific cutoffs for cardiac troponin in Denmark as well as internationally as recommended in guidelines by professional cardiological societies.

ELIGIBILITY:
Inclusion criteria for the primary cohort:

The primary cohort will include the women and men who are expected to be most significantly impacted by the intervention, and this group is specifically defined by

1. Presenting complaints suggestive of ACS
2. At least one cTn measurement within 24 hours of admission
3. A peak cTn value between the current sex-uniform manufacturer-derived 99th percentile URL and the novel sex-and population-specific 99th percentile URLs for women and men.

Presenting complaints suggestive of ACS will be identified in hospital records by the following presenting complaints of "chest pain" (DR074), "angina pectoris" (DI20) and "myocardial infarction" (DI21), "abdominal and pelvic pain" (DR10), "pain in the throat and chest" (DR07), "dyspnea" (DR060), "reflux" (DK21) and "observation due to suspicion of another cardiovascular disorder" (DZ035).

Study participants are included at their index admission, and subsequent admissions are evaluated in follow up analyses.

Exclusion criteria:

* Age < 18 years
* Patients with discharge diagnoses with conditions like pericarditis, myocarditis, endocarditis, cardiomyopathy, valve disease, arrhythmia, heart failure, pulmonary embolism, digestive system diseases, diseases of the urinary and reproductive organs, and diseases of bones, muscles, and connective tissue, and no discharge diagnosis of myocardial infarction or angina pectoris

The initial month following the implementation of the new sex-specific 99th percentile URLs will be excluded from consideration, as it will be seen as an adjustment period. Consequently, the intervention period will be extended by one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
A composite of myocardial infarction, unplanned revascularisation (after index admission) or all cause mortality within 1 year of first admission for the primary cohort. | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Primary cohort is defined as the cohort of women and men with suspected acute coronary syndrome (ACS) with at least two cTn measurements within 24 hours with a maximal cTn level between the current sex-uniform manufacturer-derived 99th percentiles of cTn and the newly defined sex-specific 99th percentiles for women and men.

SECONDARY OUTCOMES:
Number of women with coronary events in the primary cohort (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Primary cohort is defined as the cohort of women and men with suspected acute coronary syndrome (ACS) with at least two cTn measurements within 24 hours with a maximal cTn level between the current sex-uniform manufacturer-derived 99th percentiles of cTn and the newly defined sex-specific 99th percentiles for women and men.
  Coronary events are defined as the prevalence of cardiovascular death, myocardial infarction or unplanned revascularisation (after index admission) within 1 year of first admission.
Number of men with coronary events in the primary cohort (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Primary cohort is defined as the cohort of women and men with suspected acute coronary syndrome (ACS) with at least two cTn measurements within 24 hours with a maximal cTn level between the current sex-uniform manufacturer-derived 99th percentiles of cTn and the newly defined sex-specific 99th percentiles for women and men.
  Coronary events are defined as the prevalence of cardiovascular death, myocardial infarction or unplanned revascularisation (after index admission) within 1 year of first admission.
Number of women and men with coronary events in the primary cohort (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Primary cohort is defined as the cohort of women and men with suspected acute coronary syndrome (ACS) with at least two cTn measurements within 24 hours with a maximal cTn level between the current sex-uniform manufacturer-derived 99th percentiles of cTn and the newly defined sex-specific 99th percentiles for women and men.
  Coronary events are defined as the prevalence of cardiovascular death, myocardial infarction or unplanned revascularisation (after index admission) within 1 year of first admission.
Number of women diagnosed with acute MI (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of women diagnosed with acute MI | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of men diagnosed with acute MI (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of men diagnosed with acute MI | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The overall number of women and men diagnosed with acute MI (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
The overall number of women and men diagnosed with acute MI | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of women receiving unplanned revascularization (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
Number of women receiving revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
Number of men receiving unplanned revascularization (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
Number of men receiving revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
The overall number of women and men receiving unplanned revascularization (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
The overall number of women and men receiving revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  Revascularization is defined as Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting.
Number of women with all cause death (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of women with all cause death | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of men with over-all death (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of men with over-all death | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The overall number of women and men with over-all death (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
The overall number of women and men with over-all death | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of women receiving coronary angiographies or heart CT without revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of men receiving coronary angiographies or heart CT without revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The overall number of women and men receiving coronary angiographies or heart CT without revascularization | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
Number of women receiving treatment with aspirin, dual anti-platelet therapy and/or statins | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of men receiving treatment with aspirin, dual anti-platelet therapy and/or statins | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
The overall number of women and men receiving treatment with aspirin, dual anti-platelet therapy and/or statins | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
Number of women re-admitted | 12 months after index admission
  Readmission after index admission
Number of men re-admitted | 12 months after index admission
  Readmission after index admission
The overall number of women and men re-admitted | 12 months after index admission
  Readmission after index admission
Length of hospital stay for women | 30 days
  Calculated as days from date of index admission to date of discharge
Length of hospital stay for men | 30 days
  Calculated as days from date of index admission to date of discharge
Length of hospital stay for women and men | 30 days
  Calculated as days from date of index admission to date of discharge
The number of women diagnosed with myocardial injury and an event in the primary endpoint | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  The primary endpoint is a composite of myocardial infarction, unplanned revascularisation (after index admission) or all cause mortality within 1 year of index admission.
The number of men diagnosed with myocardial injury and an event in the primary endpoint | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  The primary endpoint is a composite of myocardial infarction, unplanned revascularisation (after index admission) or all cause mortality within 1 year of index admission.
The overall number of men diagnosed with myocardial injury and an event in the primary endpoint | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
  The primary endpoint is a composite of myocardial infarction, unplanned revascularisation (after index admission) or all cause mortality within 1 year of index admission.
The number of women diagnosed with myocardial injury | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The number of women diagnosed with myocardial injury (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
The number of men diagnosed with myocardial injury | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The number of men diagnosed with myocardial injury (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.
The overall number of women and men diagnosed with myocardial injury. | 12 months from index admission
  Time frame starts from beginning of index admission, defined as first admission in the study period.
The overall number of women and men diagnosed with myocardial injury (after index admission) | 12 months after index admission
  Time frame starts at discharge from the hospital from the index admission, defined as first admission in the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper K Iversen, MD, DMsc, Principal Investigator — Herlev Hospital, University Hospital of Copenhagen
Locations (22):
- Denmark (22):
  - Hospital of Southern Jutland, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bispebjerg & Frederiksberg Hospital, Bispebjerg
  - Rigshospitalet (Blegdamsvej), Copenhagen Ø
  - Sydvestjysk Sygehus, Esbjerg
  - Glostrup University Hospital, Glostrup Municipality
  - Gødstrup Regional Hospital, Gødstrup
  - Herlev & Gentofte Hospital, Herlev
  - C Torp-Pedersen, Hillerød
  - North Denmark Regional Hospital, Hjørring
  - Holbaek Sygehus, Holbæk
  - Horsens Hospital, Horsens
  - Amager & Hvidovre Hospital, Hvidovre
  - Sygehus Lillebælt (Kolding Sygehus & Vejle Sygehus), Kolding
  - Zealand University Hospital, Køge
  - Nykøbing Falster County Hospital, Nykøbing Falster
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Slagelse Sygehus, Slagelse
  - Svendborg Hospital, Svendborg
  - Central Jutland Regional Hospital (Viborg Hospital & Silkeborg Hospital), Viborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hasselbalch RB, Strandkjaer N, Kristensen J, Jorgensen N, Kock TO, Lange T, Ostrowski SR, Nissen J, Larsen MH, Vesterager Pedersen OB, Bor MV, Afzal S, Kamstrup PR, Dahl M, Hilsted L, Rode L, Jorgensen NR, Torp-Pedersen C, Bundgaard H, Iversen KK. Impact of age on cardiac troponin concentration among healthy individuals. Clin Biochem. 2025 Aug;138:110956. doi: 10.1016/j.clinbiochem.2025.110956. Epub 2025 Jun 11. PMID 40513714
- [Derived] Strandkjaer N, Jorgensen N, Hasselbalch RB, Kristensen J, Knudsen MSS, Kock TO, Lange T, Lindholm MG, Bruun NE, Holmvang L, Terkelsen CJ, Pedersen CK, Christensen MK, Lassen JF, Hilsted L, Ladefoged S, Nybo M, Bor MV, Dahl M, Hansen AB, Kamstrup PR, Bundgaard H, Torp-Pedersen C, Iversen KK. DANSPOT: A Multicenter Stepped-Wedge Cluster-Randomized Trial of the Reclassification of Acute Myocardial Infarction: Rationale and Study Design. J Am Heart Assoc. 2024 May 7;13(9):e033493. doi: 10.1161/JAHA.123.033493. Epub 2024 Apr 19. PMID 38639348